CLINICAL TRIAL: NCT07196176
Title: Registry on Electrophysiological Studies (EPS) at University Hospital Düsseldorf
Brief Title: Electrophysiological Registry Duesseldorf
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: EPS Registry
Record Dates: First submitted 2025-09-17; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation (AF); Atrial Flutter; Supraventricular Tachycardias; Ventricular Tachycardia (VT)
Keywords: atrial fibrillation; catheter ablation; cardioversion
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Tachycardia, Supraventricular; Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This registry at University Hospital Düsseldorf collects retrospective and prospective (from 2019 onward) data on patients undergoing electrophysiological studies (EPS), catheter ablation, and electrical cardioversion. The primary goal is to evaluate safety, efficacy, and clinical outcomes of these standard procedures in routine care. Data will be used for quality assurance and to identify prognostic patient- and procedure-related factors.

DETAILED DESCRIPTION:
This is a single-center observational registry including all patients treated with EPS, catheter ablation, or electrical cardioversion at the Department of Cardiology, Pneumology, and Angiology, University Hospital Düsseldorf. Retrospective data from 2011 onward and prospective data from 2015 onward are collected.

The registry systematically records demographic data, comorbidities, laboratory and imaging results, procedural details, and follow-up outcomes. Patients are routinely followed at 1, 3, 6, 12, and 24 months after the procedure. Additional follow-up may be performed by telephone interview with patients or referring physicians to improve data quality.

Primary endpoints focus on safety (peri- and postprocedural complications, late adverse events) and efficacy (recurrence of arrhythmias, need for repeat procedures, pacemaker implantation, or new medications). Secondary endpoints include hospitalization and all-cause mortality.

Participation does not alter routine diagnostic or therapeutic decisions, and no additional invasive procedures are performed. Data will be used for quality assurance and to improve understanding of prognostic factors, with the ultimate aim of optimizing future patient care.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo an electrophysiological study (EPS) or electrical cardioversion at University Hospital Düsseldorf since 2015 (retrospective cohort)
* Patients scheduled to undergo an EPS or electrical cardioversion at University Hospital Düsseldorf from 2019 onward (prospective cohort) •- Written informed consent for participation in the registry (prospective part only)

Exclusion Criteria:

* < 18 years
* Lack of written informed consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart rhythm disorders
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Periprocedural and postprocedural safety events | Up to 24 months after procedure
  All cardiovascular adverse events or complications occurring during hospitalization and late complications after discharge related to EPS, ablation, or electrical cardioversion.
Clinical efficacy outcomes | Up to 24 months after procedure
  Procedural success, recurrence of arrhythmias or symptoms, and need for repeat EPS/cardioversion, additional medication, or device implantation (e.g., pacemaker).

SECONDARY OUTCOMES:
All-cause mortality | Up to 24 months after procedure
  Death from any cause during follow-up.
All-cause hospitalization | Up to 24 months after procedure
  Any hospital admission for cardiovascular or non-cardiovascular reasons during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, MD, Study Chair — Division of Cardiology, Pulmonary Disease and Vascular Medicine at University Hospital Duesseldorf; Obaida Rana, MD, Principal Investigator — Division of Cardiology, Pulmonary Disease and Vascular Medicine at University Hospital Duesseldorf
Locations (1):
- University Hospital Duesseldorf, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No
not necessary as its a registry